CLINICAL TRIAL: NCT06458608
Title: Determining the Effect of Virtual Reality-Based Videos on Hemodialysis Symptoms, Vital Signs and Comfort in Hemodialysis Patients
Brief Title: Hemodiasis Patients Using Virtual Reality Video
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dilan aktepe coşar (Other)
Responsible Party: Sponsor-Investigator, Dilan aktepe coşar, lecture, Gümüşhane Universıty
Organization: Gümüşhane Universıty (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Hm20240001
Record Dates: First submitted 2024-06-09; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Hemodialysis; Symptoms; Virtual Reality; Comfort
Keywords: Hemodialysis, Virtual Reality Symptoms, Vital Signs, Comfort

STUDY DESIGN:
Intervention Model Description: No study could be taken as a reference due to the number of samples, the amount of error in the G*Power 3.1.9.6 program, α=0.05, and the lack of a previous study with 2 groups on the subject; With an effect size of 0.80 and the power of the targeted test being 0.80 (80%), a total of 42 patients (21 for each group) were calculated for two groups (experimental group, control group). Considering situations such as wanting to leave the study or death during the research, each group will be increased by 20% and a total of 50 patients will be included in the study, 25 patients for each group.
Masking Description: hile the patients were randomized; In order to keep the possibility of being affected by each other at a minimum level, the study was continued with the same application group in the same session group. For example; It's like working only with the robot cat group in the 08:00-12:00 session group on Mondays. In order to reduce the possibility of selection bias due to sample selection, "single-stage cluster type random sampling", which is a subtype of random sampling, was used. In addition, before the study, patients were informed about the study and their consent was obtained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group that watched virtual reality videos (Experimental): Pre-test data for all participants before treatment in the waiting room of the hemodialysis unit, "Structured Patient Introduction Form" (Annex-1), "Dialysis Symptom Index (DSI)" (Appendix 2), "Vital Signs Monitoring Form" (Appendix). 3),''Hemodialysis Comfort Scale Version II'' (Appendix 4) face to face interview for approximately 15 minutes is run as learning pre-test data. The intervention group was also given information about the use of virtual reality and the video content to be watched. Videos are transferred to virtual reality glasses and presented with the headset. After the hemodialysis treatment starts, the intervention psychologist researcher will watch 30 scan videos of approximately half an hour during the dialysis period, 2 sessions a week for 8 weeks, and a Turkey promotional short film presented by the researchers visually and audibly in VR (VR Shineco 3d).
  Interventions: Device: virtual reality glasses
- The group that is not allowed to watch virtual reality videos (Experimental): The hemodialysis patients in this group were not shown anything. Only data collection forms were administered to the patients before the study (pretest) and at the end of the study.
  Interventions: Device: virtual reality glasses

INTERVENTIONS:
Device: virtual reality glasses — virtual reality glasses

SUMMARY:
VR, with its developing technology, is a new technique used in the healthcare industry combined with cognitive technology to reduce the symptoms experienced by patients and to relieve the patient. This study investigates whether virtual tour environments created using virtual reality glasses have an effect on patients' vital signs, symptoms and comfort during the hemodialysis session. It is aimed to evaluate the effect of Virtual Reality Based Videos applied during hemodialysis treatment on Hemodialysis Symptoms, vital signs and Comfort.

DETAILED DESCRIPTION:
Hemodialysis (HD) is one of the treatment options used to regulate renal functions in the treatment of chronic renal failure. In hemodialysis, patients have to cope with many problems during the treatment process as well as the disease. In addition, patients require HD treatment, which lasts three to four hours, three times a week on average. Factors such as having to go to a dialysis center for these treatments, patients having to continue their lives depending on the machine, restriction of movements during the session, increased dependency of the patient, deterioration in their adaptation to professional and social relationships affect the patients' daily life activities and reduce their comfort. With the developing technology, virtual reality, a new technique in the healthcare industry, has begun to be used in nursing care in order to reduce the symptoms experienced by patients and to comfort the patient.

The virtual reality device removes the patient from the environment with the glasses and headphones attached to the person's head, along with the image on the screen and simultaneous sounds, and focuses his/her attention on the virtual video images. This study was planned as a randomized controlled study to evaluate the effect of virtual reality-based videos on hemodialysis symptoms and comfort in hemodialysis patients. The research was planned to be conducted with 50 hemodialysis patients. "Patient Introduction Form", "Dialysis Symptom Index (DSI)", "Vital Signs Monitoring Form", "Hemodialysis Comfort Scale Version II" will be used to collect data. After the scales were applied, patients in the experimental group were exposed to virtual reality glasses for 30 minutes, twice a week for 8 weeks. The video will be watched. At the end of 8 weeks, the scales will be applied again and compared with the initial scale results.

As a result, in line with the findings obtained from the research, the effect of virtual reality application on dialysis symptoms, vital signs and comfort during hemodialysis treatment will be determined and suggestions will be made to encourage patients to use virtual reality methods in the environments where they are treated.

ELIGIBILITY:
Inclusion Criteria:

- Voluntarily over 18 years

Exclusion Criteria:

* reluctant

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Hemodialysis Comfort Scale Version II (HDCS Version II) | 8 week
  The scale consists of a total of 26 items and a 5-point Likert type. HDCS Version II has six subscales (physical relaxation, physical comfort, psychospiritual comfort, psychospiritual transcendence, environmental transcendence, and sociocultural comfort).

SECONDARY OUTCOMES:
Dialysis Symptom Index (DSI) (Appendix 2) | 8 week
  It consists of a total of 30 items that evaluate the emotional and physical symptoms of dialysis patients and the severity of these symptoms.
Vital Signs Monitoring Form | 8 week
  It is a form in which patients' BP, respiratory rate, pulse, temperature and oxygen saturation values are measured and recorded once a week before and after the HD procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Dilan aktepe coşar, Principal Investigator — Gümüşhane Universıty
Locations (1):
- Gümüşhane Üniversitesi, Gümüşhane, Kelkit, Turkey (Türkiye)